CLINICAL TRIAL: NCT06680570
Title: Pulmonary capacıty, physıcal actıvıty Level and Headaches in Smokers and Non-smokers: ınsıghts From a unıversıty Student Cohort
Brief Title: Smoking and Health Among University Students
Acronym: SHUS
Status: Completed | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Sponsor
Other Study IDs: SFT; 2019/AP/0012 (Other Grant/Funding Number: Yalova University Scientific Research Projects Commission)
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Disease; Headache Disorders; Sedentary Behavior; Physical Activity Level
Keywords: Smoking; Headache; Students; Sedentary behavior
MeSH Terms: conditions — Lung Diseases; Headache Disorders; Sedentary Behavior; Smoking; Headache | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- smokers: Group: smokers Smokers Description: This group consists of university students who smoke regularly. Lung capacity, physical activity levels, carbon monoxide (CO) breath values and headache frequency will be measured and evaluated. This group was included in the study to examine the effect of smoking on these health parameters.
  Non-Smokers Description: This group consists of non-smoking university students. Lung capacity, physical activity levels and headache frequency of non-smokers will be measured and compared with the smoking group. This group was included to analyse the relationship between lung function and headache in non-smokers.
  Interventions: Diagnostic Test: Pulmonary Function Testing, Carbon Monoxide (CO) Breath Testing

INTERVENTIONS:
Diagnostic Test: Pulmonary Function Testing, Carbon Monoxide (CO) Breath Testing — Pulmonary Function Testing FEV1 and FVC spirometry tests used to measure lung capacity among both smoker and non-smoker students.
  Carbon Monoxide (CO) Breath Testing Measurements taken using a CO breath analyzer to assess CO levels in the smoker group.
  Physical Activity Assessment (IPAQ-SF) The International Physical Activity Questionnaire Short Form (IPAQ-SF) used to evaluate physical activity levels and sedentary behavior among students.
  Headache Impact Test (HIT-6) HIT-6 questionnaire used to assess the impact of headaches on daily life.
  Other Names: Headache Impact Test (HIT-6), Physical Activity Assessment (IPAQ-SF)

SUMMARY:
The goal of this observational study is to explore the associations between pulmonary capacity, physical activity levels, and headache occurrence in university students aged 18-30, focusing on differences between smokers and non-smokers. The main questions it aims to answer are:

Is there a relationship between pulmonary function (FEV1 and FVC measurements) and the frequency of headaches in university students? How do physical activity levels and sedentary behavior differ between smokers and non-smokers, and how do these factors correlate with headache prevalence? Researchers will compare smokers and non-smokers to see if smoking influences CO levels, sedentary behavior, and respiratory function, contributing to a higher incidence of headaches.

Participants will:

Complete pulmonary function tests using handheld spirometers to measure FEV1 and FVC.

Fill out the International Physical Activity Questionnaire (IPAQ-SF) to assess physical activity and sedentary behavior.

Use the Headache Impact Test (HIT-6) to evaluate headache impact on daily life. Provide carbon monoxide (CO) breath levels for analysis.

DETAILED DESCRIPTION:
This observational study investigates the relationships between pulmonary function, physical activity levels, and headache prevalence in university students, with a specific focus on the impacts of smoking. Conducted at Yalova University in Turkey, the study includes a diverse cohort of students aged 18-30, separated into two groups: smokers and non-smokers. By examining the physical health profiles and lifestyle behaviors of these students, the research aims to understand how smoking might affect respiratory function, activity levels, and the incidence of headaches within this population.

Objectives

The primary objectives are:

To determine whether pulmonary function (measured through FEV1 and FVC) is associated with headache occurrence and severity.

To assess the difference in sedentary behavior and physical activity levels between smokers and non-smokers and how these factors correlate with headache prevalence.

To analyze how elevated carbon monoxide (CO) levels from smoking affect respiratory capacity and contribute to headache incidence.

Methods

The study employs a cross-sectional design and utilizes several standardized tools for data collection:

Pulmonary Function Tests (PFTs): FEV1 (Forced Expiratory Volume in 1 second) and FVC (Forced Vital Capacity) values are recorded using a handheld spirometer. These tests provide an objective measure of lung capacity, which may be impacted by smoking.

International Physical Activity Questionnaire (IPAQ-SF): This validated questionnaire is used to assess physical activity levels, categorizing participants into low, moderate, or high activity levels, while also measuring sedentary behavior.

Headache Impact Test (HIT-6): This self-reported tool is administered to gauge the impact of headaches on daily life, allowing researchers to classify headache severity and its interference with student activities.

CO Breath Test: To assess smoking intensity, CO levels are measured using a breath analyzer, providing a clear, quantifiable indication of recent exposure to cigarette smoke.

Study Population and Exclusion Criteria Participants include male and female students aged 18-30 who are non-smokers or regular smokers. Exclusion criteria include individuals with pre-existing respiratory or cardiovascular conditions, recent respiratory infections, or recent surgeries. Students with diagnosed respiratory diseases (e.g., COPD, asthma) are excluded to ensure a focus on otherwise healthy individuals within the target age range.

Expected Outcomes

The study hypothesizes that:

Reduced lung function (lower FEV1 and FVC values) correlates with an increased frequency and severity of headaches, particularly among smokers.

Higher CO levels in smokers will be associated with greater headache prevalence and lower physical activity levels.

Sedentary behavior will be more common among non-smokers and may contribute to an increased incidence of headaches in this subgroup.

Significance The findings of this study are anticipated to provide valuable insights into the health impacts of smoking on young adults, particularly within the context of respiratory and neurological health. By establishing correlations between smoking, lung function, physical activity, and headaches, the study aims to inform targeted interventions for university students. Future public health initiatives may benefit from these findings by addressing sedentary behavior and smoking habits as key factors affecting the well-being of young adults in educational settings.

ELIGIBILITY:
Inclusion Criteria:

Being Yalova University students Aged between18-30 years

Exclusion Criteria:

Participants showing signs or diagnosed with respiratory conditions such as tuberculosis, post-tuberculosis lung disease, bronchial asthma, Chronic Obstructive Pulmonar Disease, or valvular heart disease were excluded

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young people
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | 10 month
  FVC spirometry tests (liters) used to measure lung capacity among both smoker and non-smoker students.
Forced Expiratory Volume in 1 second (FEV1) | 10 month
  FEV1 spirometry tests (liters) used to measure lung capacity among both smoker and non-smoker students.
Headache Impact Test (HIT-6) | 10 month
  Headache Impact Test questionnaire used to assess the impact of headaches on daily life.
Physical Activity Assessment (IPAQ-SF) | 10 month
  The International Physical Activity Questionnaire Short Form (IPAQ-SF) used to evaluate physical activity levels and sedentary behavior among students.
Carbon Monoxide (CO) Level | 10 month
  Measurement of carbon monoxide levels (Part Pers Million (ppm)) in exhaled breath to assess exposure from smoking.

CONTACTS AND LOCATIONS:
Overall Officials: asuman SALTAN, Principal Investigator — University of Yalova
Locations (1):
- asuman SALTAN, Yalova, Turkey (Türkiye)